CLINICAL TRIAL: NCT03812679
Title: Performance Evaluation of the AMIA Automated Peritoneal Dialysis (APD) Solution Generation System in Patients Using the AMIA APD Cycler
Brief Title: Performance Evaluation of the AMIA APD Solution Generation System in Patients End Stage Renal Disease (ESRD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated for business reasons not due to scientific data. Sufficient data was acquired to transition program development to other technologies
Sponsor: Vantive Health LLC (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BXU011787
Record Dates: First submitted 2019-01-04; First posted 2019-01-23 (Actual); Results first posted 2021-02-05 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: End Stage Renal Disease (ESRD)
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- AMIA APD Solution Generation System (Experimental): A simulated treatment will take place before the patient receives study treatment, during week 1 and after 4, 8 and 12 weeks of study treatment period. The dialysis solution generated by the simulated treatment will be collected from the system in the heater bag and used to evaluate the chemical composition of the final dialysis solution produced by patients using the AMIA APD Solution Generation System. Also, product water from the Water Device (pre-sterilizing filters) will be collected and tested at each visit.
  Interventions: Device: AMIA APD Solution Generation System

INTERVENTIONS:
Device: AMIA APD Solution Generation System — The AMIA APD Solution Generation System consists of the AMIA APD Cycler, Sharesource Platform, AMIA APD Concentrates, a disposable set, a bag tray, a Water Softener, and a Water Device (WD).

SUMMARY:
Peritoneal dialysis (PD) is a well-established treatment for renal failure including long-term management of end stage renal disease (ESRD) by continuous ambulatory peritoneal dialysis or automated peritoneal dialysis (APD).

Complementary therapies offer longer term survival for patients with ESRD. However, none of them are devoid of side effects and today their limitations are better understood by the nephrologist.

The AMIA APD Solution Generation System combines an updated AMIA APD Cycler with Sharesource Platform (previously cleared) with an in-home water system technology and leverages newly developed AMIA APD Concentrates.

The AMIA APD Concentrates, after dilution by the AMIA APD Solution Generation System, are indicated for adult patients in acute or chronic renal failure when non-dialytic medical therapy is judged to be inadequate.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 years or older.
2. Patient with ESRD receiving PD therapy, and who is already trained and regularly using the AMIA or HomeChoice APD Cycler with Dianeal PD Solution for at least 12 weeks.
3. Patient is receiving or willing and able to use Dianeal Low Calcium (2.5 mEq/L) PD prescriptive regimen at study treatment initiation per Investigator's assessment.
4. Patient demonstrates adequate PD therapy with clinical euvolemia as assessed by the Investigator with a total Kt/Vurea of a minimum of 1.7 within 45 days of Screening, or measured at Screening. If a total Kt/Vurea is not available within 45 days of Screening, it will be measured at Screening.
5. Investigator assesses that, with appropriate training, the patient will be able to successfully manage his/her dialysis treatments with the AMIA APD Solution Generation System.
6. Patient is available and is willing to complete training on the AMIA APD Solution Generation System.
7. Patient and home environment are deemed suitable for treatment with the AMIA APD Solution Generation System, while in the home.
8. Home electrical and water assessments meet suitability criteria for the AMIA APD Solution Generation System.
9. The patient's home has suitable wireless connection or patient is willing to allow installation of suitable wireless connection.
10. Patient and/or care partner (if participating) is able to read and understand English, and provide informed consent after an explanation of the proposed study. If the patient does not read and understand English, patient may still participate if he/she has a co-residing care partner who reads and understands English, assessed as adequate by the PI.
11. Women of childbearing potential (not menopausal or surgically sterile) must not be pregnant. Serum qualitative and quantitative pregnancy test will be done within 14 days prior to initiation of study product.

    * If qualitative serum β-hCG results are positive, repeat quantitative serum pregnancy test in 48 hours.
    * If quantitative serum β-hCG levels show clinically significant rise within 48 hours, serum progesterone level should be taken. Serum progesterone > 5 ng/mL will exclude a patient from the study.
12. Sexually active males and females agree to use a reliable means of contraception during the study and for 30 days afterwards (e.g., oral contraceptive and condom, intrauterine device and condom, or diaphragm with spermicide and condom).

Exclusion Criteria:

1. Patient with a history of PD catheter dysfunction within 12 weeks prior to study enrollment, as evaluated by the Investigator.
2. Patient who had episodes of peritonitis or exit site infection within 12 weeks prior to study enrollment.
3. Patient who has signs of impending or current infection including a cloudy dialysis effluent or dialysis white cell count > 100/ μL or > 0.1 x 109/ L (after a dwell time of at least 2 hours), with > 50% polymorphonuclear cells, and/or positive dialysis effluent culture.
4. Patient who has a severe primary immune deficiency or other condition that may mask clinical signs of peritonitis, as evaluated by the Investigator.
5. Patient with a history of repeated non-compliance with PD, therapy (e.g., a substantial number of missed clinic visits, missed treatments or a history of mismanagement of diet or medications), as evaluated by the Investigator.
6. Patient who has acute renal failure with the chance for recovery.
7. Patient who is pre-scheduled for a living donor kidney transplant within the next 6 months.
8. Patient who is not expected to live at least 6 months while maintaining PD treatment.
9. Patient who had major abdominal surgery within 6 months prior to study enrollment.
10. Patient with current abdominal hernia, as evaluated by the Investigator.
11. Patient with advanced liver or pulmonary disease, as evaluated by the Investigator.
12. Positive serology test for Hepatitis B Virus or Hepatitis C Virus infection, or aspartate transaminase or alanine aminotransferase > 3 x upper limit of normal at Screening.
13. Patient with diagnosed stage III or IV New York Heart Association (NYHA) heart failure.
14. Patient who has an active malignancy.
15. History of a clinically significant illness and/or clinically significant surgery within the past 14 days preceding the Screening Visit as determined by the Investigator.
16. Patient who is enrolled in another interventional clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Investigational Site, Jonesboro, Arkansas
  - Investigational Site, San Jose, California
  - Investigational Site, Jacksonville, Florida
  - Investigational Site, Chicago, Illinois
  - Investigational Site, Ann Arbor, Michigan
  - Investigational Site, Jackson, Mississippi
  - Investigational Site, New York, New York
  - Investigational Site, Cleveland, Ohio
  - Investigational Site, Temple, Texas
  - Investigational Site, Fitchburg, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AMIA APD Solution Generation System
Started | 22
Completed | 14
Not Completed | 8
Not completed — Adverse Event | 2
Not completed — Missed >4 consecutive therapy days | 1
Not completed — Renal transplant | 1
Not completed — Withdrawal by Subject | 1
Not completed — Termination of study | 2
Not completed — Water device replacement | 1

BASELINE CHARACTERISTICS:
Population: The Safety Set was based on the Intent-to-Treat principle and included all patients who received at least one treatment with the AMIA APD Solution Generation System and who had at least one measurement for the primary endpoint (either primary efficacy or primary safety).
Arm/Group | AMIA APD Solution Generation System
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (13.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5
  Black or African American | 7
  White | 9
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Tests Meeting Specifications for the Chemical Composition of Final Dialysis Solution by Visit
Description: The dialysis solution generated by the simulated treatment will be sampled from the heater bag, compared to the specifications of Baxter's approved low calcium Dianeal PD solution. The following 9 test methods will be analyzed: pH at 25 C, Color, 5- (hydroxymethyl)furfural (5HMF), Dextrose hydrous Assay (1.5%, 2.5% or 4.25%), Sodium Lactate Assay, Sodium Assay, Chloride Assay, Magnesium Chloride Hexahydrate (MgCl2.6H2O) Assay, and Calcium Chloride Dihydrate (CaCl2.2H2O) Assay. Measurements were collected using instruments such as meters, chromatography, etc. Data will be reported showing percentage of participants meeting specifications versus percentage of participants not meeting specification. If any one of the values falls outside the limits, then the particular test is considered NOT meeting specifications.
Time Frame: Week 1, 4, 8 and 12
Population: Safety Set used for analysis population. Also, Overall Number of Tests Analyzed (N) was captured, along with number of evaluable tests (n) for each individual timepoint.
Measure: Number; unit: Percentage of Tests
Units Other Than Participants: Tests
Arm/Group | AMIA APD Solution Generation System
Number analyzed (Participants) | 22
Number analyzed (Tests) | 71
Percentage of Tests
  Week 1 (1.5% Dextrose): Met Specifications: number analyzed (Tests) | 23
  Week 1 (1.5% Dextrose): Met Specifications | 91.3
  Week 1 (1.5% Dextrose): Did Not Meet Specifications: number analyzed (Tests) | 23
  Week 1 (1.5% Dextrose): Did Not Meet Specifications | 0
  Week 1 (1.5% Dextrose): Missing Results: number analyzed (Tests) | 23
  Week 1 (1.5% Dextrose): Missing Results | 8.7
  Week 4 (2.5% Dextrose): Met Specifications: number analyzed (Tests) | 20
  Week 4 (2.5% Dextrose): Met Specifications | 95
  Week 4 (2.5% Dextrose): Did Not Meet Specifications: number analyzed (Tests) | 20
  Week 4 (2.5% Dextrose): Did Not Meet Specifications | 0
  Week 4 (2.5% Dextrose): Missing Results: number analyzed (Tests) | 20
  Week 4 (2.5% Dextrose): Missing Results | 5
  Week 8 (4.25% Dextrose): Met Specifications: number analyzed (Tests) | 14
  Week 8 (4.25% Dextrose): Met Specifications | 85.7
  Week 8 (4.25% Dextrose): Did Not Meet Specifications: number analyzed (Tests) | 14
  Week 8 (4.25% Dextrose): Did Not Meet Specifications | 0
  Week 8 (4.25% Dextrose):Missing Results: number analyzed (Tests) | 14
  Week 8 (4.25% Dextrose):Missing Results | 14.3
  Week 12 (1.5% Dextrose): Met Specifications: number analyzed (Tests) | 14
  Week 12 (1.5% Dextrose): Met Specifications | 85.7
  Week 12 (1.5% Dextrose): Did Not Meet Specifications: number analyzed (Tests) | 14
  Week 12 (1.5% Dextrose): Did Not Meet Specifications | 0
  Week 12 (1.5% Dextrose): Missing Results: number analyzed (Tests) | 14
  Week 12 (1.5% Dextrose): Missing Results | 14.3

2. Primary Outcome: Percentage of Tests Meeting Specifications for the Microbiological and Chemical Testing of Product Water From Water Device (Pre-sterilizing Filters) by Visit
Description: Microbiological testing within <=0 CFU/mL limit for total aerobic microbial count (TAMC) and total yeast/mold count (TYMC) and <0.03 EU/mL limit for Endotoxins, and chemical parameters. Product water from the WD (pre-sterilizing filters) was collected and tested for microbiological (including endotoxin) contamination per USP <61> and USP <85> and chemical contaminants according to ISO 13959. Chemical parameters include aluminum, copper, fluoride, lead, nitrate, sulphate, zinc, calcium, magnesium, potassium, sodium, antimony, arsenic, barium, beryllium, cadmium, chromium, mercury, selenium, silver, thallium, nickel, cobalt, total chlorine. Chemical measurements were collected using instruments such as meters, chromatography, etc. Data will be reported showing percentage of participants meeting specifications versus percentage of participants not meeting specification. If any one of the values falls outside the limits, then the particular test is considered NOT meeting specifications.
Time Frame: Week 1, 4, 8 and 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Tests
Units Other Than Participants: Tests
Arm/Group | AMIA APD Solution Generation System
Number analyzed (Participants) | 22
Number analyzed (Tests) | 72
Percentage of Tests
  Week 1(Visit 1): Met Specifications: number analyzed (Tests) | 24
  Week 1(Visit 1): Met Specifications | 37.5
  Week 1(Visit 1): Did Not Meet Specifications: number analyzed (Tests) | 24
  Week 1(Visit 1): Did Not Meet Specifications | 0
  Week 1(Visit 1): Missing Results: number analyzed (Tests) | 24
  Week 1(Visit 1): Missing Results | 62.5
  Week 4 (Visit 2): Met Specifications: number analyzed (Tests) | 20
  Week 4 (Visit 2): Met Specifications | 60
  Week 4 (Visit 2): Did Not Meet Specifications: number analyzed (Tests) | 20
  Week 4 (Visit 2): Did Not Meet Specifications | 15
  Week 4 (Visit 2): Missing Results: number analyzed (Tests) | 20
  Week 4 (Visit 2): Missing Results | 25
  Week 8 (Visit 3): Met Specifications: number analyzed (Tests) | 14
  Week 8 (Visit 3): Met Specifications | 78.6
  Week 8 (Visit 3): Did Not Meet Specifications: number analyzed (Tests) | 14
  Week 8 (Visit 3): Did Not Meet Specifications | 7.1
  Week 8 (Visit 3): Missing Results: number analyzed (Tests) | 14
  Week 8 (Visit 3): Missing Results | 14.3
  Week 12 (Visit 4): Met Specifications: number analyzed (Tests) | 14
  Week 12 (Visit 4): Met Specifications | 64.3
  Week 12 (Visit 4): Did Not Meet Specifications: number analyzed (Tests) | 14
  Week 12 (Visit 4): Did Not Meet Specifications | 14.3
  Week 12 (Visit 4): Missing Results: number analyzed (Tests) | 14
  Week 12 (Visit 4): Missing Results | 21.4

3. Primary Outcome: Percentage of Tests Meeting Specifications for the Microbiological Testing of Product Water From Holding Bag (Post-sterilizing Filters) by Visit
Description: Microbiological testing within <=0 CFU/mL limit for TAMC and TYMC and <0.03 EU/mL limit for Endotoxins. Data will be reported showing percentage of participants meeting specifications versus percentage of participants not meeting specification. If any one of the values falls outside the limits, then the particular test is considered NOT meeting specifications. A test was considered as meeting specifications if all of the following parameters fell within the specified limits: tryptic soy broth growth, fluid thioglycolate growth, and endotoxins. Water in the holding bag was collected and tested for microbiological contamination and endotoxin levels per USP <71> and USP <85>.
Time Frame: Week 1, 4, 8 and 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Tests
Units Other Than Participants: Tests
Arm/Group | AMIA APD Solution Generation System
Number analyzed (Participants) | 22
Number analyzed (Tests) | 71
Percentage of Tests
  Week 1 (Visit 1): Met Specifications: number analyzed (Tests) | 23
  Week 1 (Visit 1): Met Specifications | 100
  Week 1 (Visit 1): Did Not Meet Specifications: number analyzed (Tests) | 23
  Week 1 (Visit 1): Did Not Meet Specifications | 0
  Week 1 (Visit 1): Missing Results: number analyzed (Tests) | 23
  Week 1 (Visit 1): Missing Results | 0
  Week 4 (Visit 2): Met Specifications: number analyzed (Tests) | 20
  Week 4 (Visit 2): Met Specifications | 100
  Week 4 (Visit 2): Did Not Meet Specifications: number analyzed (Tests) | 20
  Week 4 (Visit 2): Did Not Meet Specifications | 0
  Week 4 (Visit 2): Missing Results: number analyzed (Tests) | 20
  Week 4 (Visit 2): Missing Results | 0
  Week 8 (Visit 3): Met Specifications: number analyzed (Tests) | 14
  Week 8 (Visit 3): Met Specifications | 92.9
  Week 8 (Visit 3): Did Not Meet Specifications: number analyzed (Tests) | 14
  Week 8 (Visit 3): Did Not Meet Specifications | 0
  Week 8 (Visit 3): Missing Results: number analyzed (Tests) | 14
  Week 8 (Visit 3): Missing Results | 7.1
  Week 12 (Visit 4): Met Specifications: number analyzed (Tests) | 14
  Week 12 (Visit 4): Met Specifications | 85.7
  Week 12 (Visit 4): Did Not Meet Specifications: number analyzed (Tests) | 14
  Week 12 (Visit 4): Did Not Meet Specifications | 0
  Week 12 (Visit 4): Missing Results: number analyzed (Tests) | 14
  Week 12 (Visit 4): Missing Results | 14.3

4. Secondary Outcome: Change From Baseline in Total Kt/Vurea at Week 5, 6, 7, or 8
Description: Peritoneal dialysis adequacy will be measured by sample collection and calculation of Total Kt/Vurea. Weekly peritoneal Kt/Vurea was calculated from blood and 24-hour PD effluent samples and renal Kt/Vurea was calculated from 24-hour collection of urine samples (if applicable) and blood samples after the patient had been dialyzing with the AMIA APD Solution Generation System for at least 4 weeks. Total Kt/Vurea is the sum of peritoneal Kt/Vurea and renal Kt/Vurea. Note: This secondary efficacy endpoint was measured by sample collection and calculation of total Kt/Vurea, occurring one time during Week 5, 6, 7, or 8 of the Study Treatment Period.
Time Frame: Baseline, Week 5 or Week 6 or Week 7 or Week 8
Population: Safety Set
Measure: Mean (Standard Deviation); unit: Kt/Vurea
Arm/Group | AMIA APD Solution Generation System
Number analyzed (Participants) | 15
Kt/Vurea | -0.15 (0.370)

ADVERSE EVENTS:
Time Frame: AEs and SAEs will be collected after the informed consent is signed and will continue to be collected throughout the Study Treatment Period and during the follow-up period of 5 days after the last study treatment.
Arm/Group | AMIA APD Solution Generation System
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 3/22
Other Adverse Events (participants affected / at risk) | 2/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMIA APD Solution Generation System (N=22)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMIA APD Solution Generation System (N=22)
Hypotension (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The study was terminated for business reasons not due to scientific data. Sufficient data was acquired to transition program development to other technologies. All enrolled subjects had completed treatment at the time that the US was impacted by COVID-19.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor reserves the right of prior review and approval of data from this study relative to the potential release of proprietary information to any publication or for any presentation.

DOCUMENTS (2):
  • Study Protocol (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT03812679/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/79/NCT03812679/SAP_001.pdf